CLINICAL TRIAL: NCT04451304
Title: Cardiorespiratory Autonomic Reflexes During Superselective Ophthalmic Artery Chemotherapy for Retinoblastoma in Children: a Prospective Observational Study.
Brief Title: Autonomic Reflexes During Intra-arterial Chemotherapy for Retinoblastoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mariana Fontes Lima Neville, Principal Investigator, Federal University of São Paulo
Other Study IDs: CAAE 28598120.5.0000.5505
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Retinoblastoma; Retinoblastoma Bilateral; Chemotherapy Effect
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective observational study in patients undergoing intra-arterial ophthalmic artery chemotherapy for the treatment of retinoblastoma. The main objective of the study is to evaluate the incidence of cardiorespiratory autonomic reflexes in these patients and to investigate the association between autonomic reflexes and perioperative clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with retinoblastoma and submitted to intra-arterial chemotherapy during the study period
* Informed consent form signed and dated by legal guardian and investigator
* Informed assent form signed by the patient if appropriate

Exclusion Criteria:

* Refusal of the patient or guardian to participate in the research project

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing cancer treatment for unilateral or bilateral retinoblastoma at the Instituto de Oncologia Pediátrica da Universidade Federal de São Paulo - GRAACC, São Paulo - Brasil.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory autonomic reflexes incidence | from the admission of the patient in the operating room until the end of the procedure (intra-arterial chemotherapy)
  To evaluate the incidence of cardiorespiratory autonomic reflexes during intra-arterial chemotherapy of the ophthalmic artery in a child cancer center.

SECONDARY OUTCOMES:
Clinical background and autonomic reflexes occurence | from the admission of the patient in the operating room until the end of the procedure.
  To evaluate the association between perioperative characteristics (both baseline and intraoperative characteristics) and the incidence of cardiorespiratory autonomic reflexes

CONTACTS AND LOCATIONS:
Overall Officials: Mariana F Lima, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil